CLINICAL TRIAL: NCT00767390
Title: CARTO 3 ACL Patches Effectiveness Over Prolonged Clinical Case
Brief Title: CARTO 3 Human Patch Study
Acronym: Human Patch
Status: Withdrawn | Type: Observational
Why Stopped: The required results were obtained through alternate methodology
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Rep2952
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: ACL Patch Placement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACL Patch
  Interventions: Device: ACL Patch

INTERVENTIONS:
Device: ACL Patch — Observe and characterize the changes in relative conductivity between the six ACL patches over period of six hours. Investigation only involves passive data collection on pressure impact and adhesiveness properties of ACL patches.

SUMMARY:
The Purpose of this clinical investigation is to observe the changes in relative conductivity between the six ACL patches over time. In addition, the clinical investigation will evaluate the impact of prolonged placement of the ACL patches on subjects' skin on the chest and back. During the study the adhesiveness properties of the patches will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Signed Subject Informed Consent Form
* Healthy subject
* Age Range: 20 - 50 years
* BMI - half o the subjects 18-25 and half >25
* Chest cage normal anatomy and dimensions
* No history of skin contact patch allergy, of any kind

Exclusion Criteria:

* Chest cage bony deformity
* Known skin allergies to patches, or dermatological conditions requiring therapy
* Presence of any active skin lesion on chest or back
* Any condition that preclude subject from lying down for six hours with minimal movement
* Pregnancy
* Subjects with devices, such as pace makers, IC, loop recorder

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10

PRIMARY OUTCOMES:
Absence of any clinically significant trauma to skin of the subjects at the ACL patches placement sites. | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Giris Jacob, M.D., Principal Investigator — Rambam Health Care Campus